CLINICAL TRIAL: NCT05821413
Title: Implementation, Evaluation, and Cost Effectiveness of a Data-to-Care Strategy to Improve HIV Continuum Outcomes for Out of Care PLWH in Ukraine
Brief Title: Implementation a Data-to-Care Strategy to Improve HIV Continuum Outcomes for Out of Care People Living With HIV (PLWH) in Ukraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Ukrainian Institute on Public Health Policy (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 00018465; R34DA053143 (NIH); IRB00018465 (Other: JHSPH IRB)
Record Dates: First submitted 2023-04-07; First posted 2023-04-20 (Actual); Results first posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Data to Care (Experimental): Clinics randomized to the intervention arm will implement the data to care strategy, which includes a 5-step process: (1) identify not-in-care PLWH using the a medical information system, (2) verify eligibility criteria, (3) contact patients and invite to visit the clinic, (4) determine care status and reengage into care, and (5) provide case management services and confirm engagement in care.
  Interventions: Behavioral: Data to care
- Standard of Care (Active Comparator): Participants in the standard of care sites will receive existing case management and supportive services from the HIV clinic.
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Data to care — Participants meet with a case manager who asks about health, basic needs such as housing and finances, and relationships and support systems. A score is assigned that reflects how much support is needed. A care plan is developed to address areas of need. The case manager meets regularly with participants to determine if needs are being met and identify strategies for meeting those needs. Participants with higher scores will receive more intensive contact with case managers, typically every month, until their level of need goes down. All participants will have their level and types of needs reassessed to determine if they need additional support or are moving toward self-management. Participants work with case managers for 6 months.
  Arms: Data to Care
Behavioral: Standard of Care — Participants can use standard case management and other services offered by the clinic.
  Arms: Standard of Care

SUMMARY:
The goal of this clinical trial is to study the preliminary effectiveness of a data to care intervention versus standard of care for people living with HIV in Ukraine. The main questions it aims to answer are:

* Does a data to care strategy improve primary outcomes of HIV care engagement, antiretroviral therapy initiation or re-initiation, and viral suppression among not-in-care people living with HIV?
* Does a data to care strategy improve secondary outcomes of engagement or re-engagement in ancillary services (e.g., drug treatment) and quality of life?

DETAILED DESCRIPTION:
The goal of this project is to develop and pilot a data-to-care strategy to improve HIV care outcomes among HIV-positive people who inject drugs (PWID) in Ukraine. Data-to-Care (D2C) is a high-impact public health strategy that integrates multiple sources of data such as clinical data from medical information systems, surveillance data, and ongoing case management assessments with clients to identify people living with HIV (PLWH) who are not in care, engage the participants in care, and manage the HIV Care Continuum. D2C strategies complement evidence-based practices for HIV care adherence by integrating clinical and case management data at multiple points along the HIV care continuum, using systematic assessments to identify unmet needs such as substance abuse treatment and make appropriate care referrals, and using data to inform practice changes and improve linkage to and retention in care. D2C strategies have been effectively implemented in jurisdictions throughout the United States but are not standard of care in low- and middle-income countries (LMICs) such as Ukraine. In Ukraine, of the approximately 250,000 estimated people living with HIV in Ukraine, only 44% are receiving antiretroviral therapy (ART). At least 50% of PLWH in Ukraine acquired HIV though intravenous drug use and are likely to be active PWID. ART use rates are particularly low among HIV-positive PWID, with only 38% on ART and 28% virally suppressed. This study's Specific Aims are: (1) to adapt a D2C implementation strategy for Ukraine; (2) to study preliminary effectiveness of a D2C strategy versus standard of care on primary outcomes of HIV care engagement, ART initiation or re-initiation, and viral suppression among not-in-care PWID living with HIV (n=160);and (3) to assess the feasibility, acceptability, implementation-related processes and costs of the D2C strategy. This study will use a cluster randomized control trial in high priority regions in Ukraine (4 clinical settings and 160 total participants). Outcomes will be assessed at 6 and 12- months post-baseline. Ukraine is well-positioned as a site to identify how D2C strategies can be implemented in LMICs. With the support of international stakeholders, the Ukrainian Ministry of Health is actively promoting the use of a medical information system (MIS) at the HIV clinic level. The MIS contains patient-level information on HIV care appointments kept, medication prescriptions, all diagnosed co-morbidities, and clinical and laboratory test results. This information can be mobilized in a D2C strategy that tracks patients through the care continuum, uses data to make decisions about patient care and improve case management practices, attends to psychosocial factors that affect medication adherence (e.g., mental health, addiction), and coordinates the provision of non-clinical social services. This project seeks to develop and test an intervention that influence organizational structure, climate, and culture to promote dissemination and adoption of evidence-based practices; and evaluate the adaptation process, and subsequent effectiveness of evidence-based interventions when implemented in real-world settings.

ELIGIBILITY:
Inclusion Criteria:

* Registered in the Ukrainian Medical Information System as having received an HIV diagnosis at any time in the past
* missed a clinical visit (medication pick-up or other) more than 7 days ago
* registered with injection drug use (IDU) as probable mode of HIV transmission, or history of IDU documented at any clinical visit
* not been contacted by other clinical staff after the current missed visit
* 18 years or older

Exclusion Criteria:

* Patient is already re-engaged in care and visited the clinic recently
* Patient has sufficient supply of medications (available to him for any reason)
* Patient moved to another clinic, city, country, or penitentiary institution

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2023-06-16 (Actual); Primary Completion 2024-11-13 (Actual); Study Completion 2024-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill Owczarzak, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Ukrainian Institute on Public Health Policy, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place between June and October 2023 at four specialized HIV care clinics in Ukraine (Dnipro, Odesa, Kyiv, Poltava). Eligible patient lists were generated and randomly sorted at each site. Outreach specialists contacted patients sequentially in the order they appeared and conducted brief scripted counseling to encourage them to visit the clinic, mentioning the opportunity to enroll in the study.
Pre-assignment Details: Sites were randomized prior to participant recruitment.
Units Other Than Participants: Clinics
Groups:
- Data to Care: Two clinics randomized to the intervention arm will implement the data to care strategy, which includes a 5-step process: (1) identify not-in-care PLWH using the a medical information system, (2) verify eligibility criteria, (3) contact patients and invite to visit the clinic, (4) determine care status and reengage into care, and (5) provide case management services and confirm engagement in care.
- Standard of Care: Participants in the two standard of care sites will receive existing case management and supportive services from the HIV clinic.
Period: Overall Study
Arm/Group | Data to Care | Standard of Care
Started | 80; 2 Clinics | 80; 2 Clinics
Completed | 80; 2 Clinics | 80; 2 Clinics
Not Completed | 0; 0 Clinics | 0; 0 Clinics

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Data to Care | Standard of Care | Total
Number analyzed (Participants) | 80 | 80 | 160
Age, Customized [Count of Participants; unit: Participants]
  18 to 40 years of age | 29 | 20 | 49
  41 to 50 years of age | 33 | 44 | 77
  51 or older years of age | 18 | 16 | 34
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 30 | 53
  Male | 57 | 50 | 107
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Engaged in HIV Care as Assessed by Number of Clinical Visits
Description: At least 3 clinical visits with at least 3 months apart within 12 months after study enrollment
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Data to Care | Standard of Care
Number analyzed (Participants) | 80 | 80
Participants | 34 | 58
Statistical Analysis 1: Comparison: Data to Care vs Standard of Care; Test type: Superiority; p < .001, Fisher Exact

2. Primary Outcome: Number of Participants Initiating ART (re-)Initiation
Description: Initiating or re-initiating ART within 3 months after study enrollment
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Data to Care | Standard of Care
Number analyzed (Participants) | 80 | 80
Participants | 80 | 78
Statistical Analysis 1: Comparison: Data to Care vs Standard of Care; Test type: Superiority; p = .50, Fisher Exact

3. Primary Outcome: Number of Participants ART Adherent as Assessed by the Percentage of Days in Possession of Medication
Description: Number of participants ART adherent assessed by the percentage of days in possession of medication (pharmacy refill gap method)
Time Frame: One month
Measure: Count of Participants; unit: Participants
Arm/Group | Data to Care | Standard of Care
Number analyzed (Participants) | 80 | 80
Participants | 64 | 40
Statistical Analysis 1: Comparison: Data to Care vs Standard of Care; Test type: Superiority; p < .001, Fisher Exact

4. Primary Outcome: Number of Participants With HIV Viral Suppression as Assessed by Viral Load (VL) Test
Description: Having at least one VL test with <200cp/ml and none with >=200cp/ml within 12 months after study enrollment
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Data to Care | Standard of Care
Number analyzed (Participants) | 80 | 80
Participants | 57 | 54
Statistical Analysis 1: Comparison: Data to Care vs Standard of Care; Test type: Superiority; p = .73, Fisher Exact

5. Secondary Outcome: Number of Participants With Substantial or Severe Substance Use as Assessed by the Drug Abuse Screening Test (DAST-10)
Description: The Drug Abuse Screening Test (DAST-10) is a 10-item brief screening tool. Each question requires a yes or no response. This tool assesses drug use, not including alcohol or tobacco use. Scores of 0 indicates no problems; 1-2 indicates low level, 3-5 indicates moderate level, 6-8 indicates substantial level, and 9-10 is severe.
Time Frame: 6 months
Population: Participants with data collected
Measure: Count of Participants; unit: Participants
Arm/Group | Data to Care | Standard of Care
Number analyzed (Participants) | 71 | 74
Participants | 13 | 33
Statistical Analysis 1: Comparison: Data to Care vs Standard of Care; Test type: Superiority; p < .001, Fisher Exact

6. Secondary Outcome: Number of Participants With Moderate or Severe Depressive Symptoms as Assessed by the Patient Health Questionnaire (PHQ-9)
Description: The Patient Health Questionnaire (PHQ-9) assesses degree of depression severity. Total scores of 5, 10, 15, and 20 represent cutpoints for mild, moderate, moderately severe and severe depression, respectively. The PHQ-9 scores range from 0-27. Scores of 10 or higher are indicative of moderate or severe depressive symptoms.
Time Frame: 6 months
Population: Participants with data collected
Measure: Count of Participants; unit: Participants
Arm/Group | Data to Care | Standard of Care
Number analyzed (Participants) | 79 | 78
Participants | 15 | 20
Statistical Analysis 1: Comparison: Data to Care vs Standard of Care; Test type: Superiority; p = .34, Fisher Exact

7. Secondary Outcome: Health-Related Quality of Life as Assessed by SF12
Description: General Health Function as measured by the Physical Component of the Medical Outcomes Study SF-12. The t-scores are based on a standardized reference population with m = 50 and SD = 10. Higher scores indicate higher functioning.
Time Frame: 6 months
Population: Participants with data collected
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | Data to Care | Standard of Care
Number analyzed (Participants) | 71 | 74
t-score | 48.5 (8.4) | 43.8 (8.8)
Statistical Analysis 1: Comparison: Data to Care vs Standard of Care; Test type: Superiority; p = .001, t-test, 2 sided

8. Secondary Outcome: HIV-related Risk Behaviors
Description: HIV transmission risk score based on self-reported episodes of sexual intercourse. The score is the expected number of onward HIV transmissions over one year (X10000) estimated from Bernoulli transmission models. Higher scores indicate higher risk of onward HIV transmission. The index does not have an upper limit. The Lower limit is 0, and the observed range is 0 - 158.8.
Time Frame: 6 months
Population: Participants with data collected
Measure: Median (Inter-Quartile Range); unit: risk score
Arm/Group | Data to Care | Standard of Care
Number analyzed (Participants) | 71 | 74
risk score | 0 [0 to 4.0] | 0 [0 to 3.2]
Statistical Analysis 1: Comparison: Data to Care vs Standard of Care; Test type: Superiority; p = .57, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Trust in Physicians as Assessed by the Trust in Physician Scale (TPS)
Description: Assesses beliefs, opinions, and attitudes about doctors and health issues. The Trust in Physician Scale is an 11-item self-report instrument developed to assess an individual's trust in his/her physician. The items use a five point scale (1=Strongly Disagree to 5= Strongly Agree), and the scale has a possible range of 11-55 with higher scores indicating higher trust in physicians.
Time Frame: One Year
Population: Participants with data collected
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Data to Care | Standard of Care
Number analyzed (Participants) | 71 | 74
score on a scale | 39.2 (7.6) | 38.5 (5.3)
Statistical Analysis 1: Comparison: Data to Care vs Standard of Care; Test type: Superiority; p = .64, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: From enrollment to 12 months post-enrollment
Arm/Group | Data to Care | Standard of Care
All-Cause Mortality (participants affected / at risk) | 2/80 | 5/80
Serious Adverse Events (participants affected / at risk) | 2/80 | 5/80
Other Adverse Events (participants affected / at risk) | 1/80 | 5/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Data to Care (N=80) | Standard of Care (N=80)
Mortality due to drug overdose (Injury, poisoning and procedural complications) | 1 | 1 — Drug overdose
Mortality due to bacterial pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Death due to primary thrombophilia (Blood and lymphatic system disorders) | 0 | 1
Mortality due to stroke (Nervous system disorders) | 1 | 0
Mortality due to undetermined cause (General disorders) | 0 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Data to Care (N=80) | Standard of Care (N=80)
Suicidal ideation (Psychiatric disorders) | 1 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-21): https://cdn.clinicaltrials.gov/large-docs/13/NCT05821413/Prot_SAP_000.pdf
  • Informed Consent Form (2023-03-21): https://cdn.clinicaltrials.gov/large-docs/13/NCT05821413/ICF_001.pdf